CLINICAL TRIAL: NCT07381712
Title: High-Flow Nasal Cannula Versus Non-Invasive Ventilation for Acute Respiratory Failure in Pulmonary Embolism: A Randomized Controlled Trial on Weaning Success and Survival"
Brief Title: High-Flow Nasal Cannula Versus Non-Invasive Ventilation for Acute Respiratory Failure in Pulmonary Embolism.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Montaser Gamal Ahmed, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HFNCvs NIV in PE
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Embolism
Keywords: NIV,HFNC
MeSH Terms: conditions — Pulmonary Embolism | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC group (Experimental): Included patients in this arm will exposed to HFNC as a modality for ventilatory support for patients with pulmonary embolism admitted to RICU.
  Interventions: Device: High-Flow Nasal Cannula (HFNC)
- NIV group (Experimental): Included patients in this arm will exposed to NIV as a modality for ventilatory support for patients with pulmonary embolism admitted to RICU.
  Interventions: Device: Non-Invasive Ventilation (NIV)

INTERVENTIONS:
Device: High-Flow Nasal Cannula (HFNC) — Patients randomized to the HFNC arm will receive heated, humidified oxygen at flow rates up to 60 L/min, with FiO₂ titrated to maintain SpO₂ within the target range (92-96%).
  Arms: HFNC group
Device: Non-Invasive Ventilation (NIV) — In the NIV arm, BiPAP devices will be used with an oronasal mask interface, adjusting inspiratory and expiratory pressures according to patient tolerance and ABG results.
  Arms: NIV group

SUMMARY:
Acute pulmonary embolism (PE) often causes hypoxemic respiratory failure through ventilation-perfusion mismatch and right-ventricular (RV) strain; supportive oxygenation plus prompt anticoagulation are crucial to care . Current guidelines advise supplemental oxygen and escalation according to hemodynamic/respiratory status, but do not identify an optimal noninvasive modality for PE-related respiratory failure.

DETAILED DESCRIPTION:
Acute pulmonary embolism (PE) often causes hypoxemic respiratory failure through ventilation-perfusion mismatch and right-ventricular (RV) strain; supportive oxygenation plus prompt anticoagulation are crucial to care . Current guidelines advise supplemental oxygen and escalation according to hemodynamic/respiratory status, but do not identify an optimal noninvasive modality for PE-related respiratory failure .. Non-invasive ventilation (NIV) can correct hypoxemia, yet applied positive pressure may adversely affect RV preload/afterload in PE and is frequently limited by intolerance . High-flow nasal cannula (HFNC) provides heated, humidified flows up to 60 L/min, improves oxygenation, reduces work of breathing, and enhances comfort versus conventional oxygen; in general hypoxemic acute respiratory failure (AHRF), HFNC reduced escalation and intubation compared with standard oxygen and, in some analyses, performed at least as well as NIV . Evidence specific to PE is emerging: a retrospective cohort and case series reported rapid improvements in oxygenation and respiratory distress with HFNC, with good tolerance and no major hemodynamic compromise. By avoiding mask-related intolerance and reducing harmful intrathoracic pressure effects while delivering consistent high FiO₂ and modest PEEP, HFNC may facilitate faster de-escalation and better outcomes than NIV in PE-related AHRF, a population for whom definitive comparative trials are lacking.

ELIGIBILITY:
Inclusion Criteria:

- 1. Age ≥18 y; presented with acute PE confirmed by CTPA or high-probability V/Q.

2. AHRF needing non-invasive support; provided that patients able to protect airway and hemodynamically stable without escalating vasopressors

Exclusion Criteria:

* 1. Immediate indication for intubation; high-risk (massive) PE with shock requiring advanced airway/vasopressors; active major bleeding; untreated pneumothorax.

  2. Contraindications/intolerance to assigned modality (e.g., facial trauma for NIV; complete nasal obstruction for HFNC).

  3. Do-Not-Intubate orders; pregnancy ; concomitant respiratory failure primarily due to another process requiring a different pathway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Weaning success at 48 h | 48 hours
  the ability of the patient to maintain spontaneous breathing without the need for reintubation, escalation to invasive mechanical ventilation, or initiation of rescue non-invasive ventilation within 48 hours. Patients who remained clinically stable, with acceptable gas exchange and no signs of respiratory failure during this period, were considered to have achieved weaning success.

CONTACTS AND LOCATIONS:
Overall Officials: montaser G ahmed, phD, Principal Investigator — Department of Chest Diseases, Assiut University Hospitals, Egypt
Locations (1):
- Assiut University Hospitals, Asyut, أسيوط - Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No